CLINICAL TRIAL: NCT03883685
Title: The Effect of Probiotics on Obesity. Metabolic Endotoxemia and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Collaborators: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Sondos Harfil, lecturer, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC-18-05-23-01
Record Dates: First submitted 2019-03-11; First posted 2019-03-21 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: both drugs pills and placebo pills are provided in identical pharmaceutical shape and packing, and provided by the same manufacturer. Participants is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 40 subjects will be randomly allocated to receive probiotics pills for consecutive 8 weeks.
  Interventions: Dietary Supplement: Probiotane
- Control group (Placebo Comparator): 40 subjects will be randomly allocated to receive placebo pills for consecutive 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotane — probiotics capsules of blended strains including Lactobacillus acidophilus, L. casei and L. rhamnosus
  Arms: experimental group
Dietary Supplement: Placebo — Placebo
  Arms: Control group

SUMMARY:
In spite of the growing evidence for the beneficial effects of probiotics, their anti-obesity effects are not well examined. No previous studies were conducted in this research area in the UAE. Hence, the aims of this study are to 1) Investigate the link between metabolic derangements associated with obesity and levels of LPS and LBP; 2) Study the relatedness of low grade inflammation with the ME; 3) Investigate the food intake assessment; and 4) Investigate the effectiveness of probiotics supplement on the obesity, ME and inflammation.

This project will have two phases: 1) a cross-sectional, in which 250 adults will be recruited for the collection of anthropometric measures, food intake, and fasting blood samples to measure serum LPS, LBP, Lipid profile, IR, insulin-like growth factor, hs-CRP, IL-6, and glucose. 2) Intervention phase, in which 50 overweight subjects will be randomly assigned to either receive a daily probiotic (25 subjects) or a placebo capsule (25 subjects) during the intervention period.

DETAILED DESCRIPTION:
General Objective:

To study the relatedness of obesity, with the associated metabolic endotoxemia and low-grade inflammation, and the effectiveness of probiotics intervention in adults, in UAE.

Specific Aims:

* Investigate the link between metabolic derangements associated with obesity and levels of LPS and LBP among the population in Sharjah, UAE.
* To examine the associated factors of obesity among the same population, including socio-demographic data, anthropometric measures, body composition analysis, and food frequency assessment.
* To investigate the correlation of the inflammatory marker Il-6 and hs-CRP to the levels of endotoxemia in lean, overweight and obese subjects.
* To evaluate the change in endotoxemia, body mass index (BMI) and inflammatory markers, after consumption of probiotics capsules of blended strains of Lactobacillus for 8 consecutive weeks among overweight and obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Accepts healthy volunteers
* 250 male and female
* age (18 - 55 yrs.)
* living in Dubai or Sharjah.

Exclusion Criteria:

* Pregnant breastfeeding or post menopause female
* individuals with thyroid
* individuals with liver, kidney or internal organs disorders
* individuals with signs of hypersensitivity
* individuals with have known allergy to probiotics, immune-disorder, malignant tumor.
* individuals with any major surgery during the last 6 months
* current smokers individuals with, acute illness within 2 weeks before collecting blood samples

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
80 participants characterized with obesity will be assessed for endotoxemia using LAL Chromogenic Endpoint Assay | 8 weeks
  Estimate the serum levels of LPS (EU/ml) before and after intervention period.
80 participants characterized with obesity will be assessed for body mass index (BMI) before and after the intervention period | 8 weeks
  BMI ( kg/m2)
Lipopolysacharide binding protein (LBP) will be assessed in the participants before and after intervention period. | 8 weeks
  LBP plasma level (ng/ml) will be assayed using ELISA technique
IL-6 serum will be assessed in participants before and after the intervention. | 8 weeks
  IL-6 serum will be assayed using ELISA
hs-CRP serum level will be assessed in participants before and after the intervention | 8 weeke
  hs-CRP will be assayed using immunoturbidimetry (ITM)
TNF-alpha serum level will be assessed in participants before and after the intervention | 8 weeks
  TNF-alpha will be assayed using ELISA technique
Lipid profile will be assayed for all participants before and after the intervention | 8 weeks
  measurement of serum levels of TG, HDL,LDL,

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Raed AbuOdeh, PhD, Study Chair — University of Sharjah
Locations (1):
- Sondos Harfil, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
All information and data will be shared with Dr. Raed AbuOdeh and all the coinvestigators
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All information will be available during and after the completion of the study for one year.
Access Criteria: Soft copy